CLINICAL TRIAL: NCT06483828
Title: The Impact of Dental Anxiety Coping Module on Children with Dental Anxiety: a Randomised Controlled Trial
Brief Title: Impact of Dental Anxiety Coping Module on Children with Dental Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DF CD 2405/0011 (P)
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-06

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Baseline MY-ACDAS and HRV-Biofeedback assessment followed with dental procedures (dental charting and oral prophylaxis). HRV-Biofeedback will be recorded during dental procedures. Once completed, post dental procedures assessment of MY-ACDAS and HRV-Biofeedback will be recorded.
- Intervention group (Experimental): Baseline MY-ACDAS and HRV-Biofeedback assessment followed Dental Anxiety Coping Module. The participants will continue with dental procedures (dental charting and oral prophylaxis). HRV-Biofeedback will be recorded during dental procedures. Once completed, post dental procedures assessment of MY-ACDAS and HRV-Biofeedback will be recorded.
  Interventions: Behavioral: Dental Anxiety Coping Module

INTERVENTIONS:
Behavioral: Dental Anxiety Coping Module — Dental tour where participants will be introduced to the dental clinic setting while Expressive Art Therapy, participants will engage with activity of making collage and finger painting.
  Arms: Intervention group

SUMMARY:
The aim of this study is to evaluate the impact of the Dental Anxiety Coping Module (DACM) in children with dental anxiety. The main questions to answer are:

1. Will the Dental Anxiety Coping Module has any effect on dental anxiety in primary school children based on MY-ACDAS and HRV-Biofeedback?
2. Is there any difference in dental anxiety between control and intervention group on baseline and post-test measured with MY-ACDAS?
3. Is there any difference in dental anxiety between control and intervention group on baseline, during and post-test measured with and HRV-Biofeedback?

DETAILED DESCRIPTION:
Dental Anxiety Coping Module (DACM) is a combination of Dental Tour and Expressive Art Therapy. Participants will be randomised into 2 groups, Control group and Intervention group (with DACM). Control group will have dental procedure without any intervention. While the Intervention group will start with dental tour where they will be shown around the dental clinic followed by Expressive Art Therapy where they will have collage and finger painting done. After DACM, participants will continue with the same dental procedure as the control group.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian child, age 7 to 11 years old that understand basic Malay and English language.
* Children that fulfil both MY-ACDAS score 26 and above and HRV-Biofeedback of very low coherence score (incoherence).
* Children with American Society of Anaesthesiologists (ASA) I and ASA II classification.

Exclusion Criteria:

* Children requiring emergency treatment such as pain, facial cellulitis, and trauma cases.
* Child with learning disabilities, hearing, or visual impairment, developmental or intellectual disability and cognitive impairment.
* Parents/guardians who refuse to allow their child to participate in this trial.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-04 (Estimated); Study Completion 2025-08-04 (Estimated)

PRIMARY OUTCOMES:
Changes in Malaysian- Abeer Children Dental Anxiety Scale (MY-ACDAS) score | Before intervention and dental procedure and immediately afterwards on the same day
  Malaysian- Abeer Children Dental Anxiety Scale (MY-ACDAS) range value from 13-39, a child is considered anxious if his/her overall score is equal or more than 26. Hence participant that score 26 and above considered having dental anxiety and will be included in the study

SECONDARY OUTCOMES:
Changes in HRV-Biofeedback coherence | Before intervention and dental procedure, during dental procedure and immediately afterwards on the same day
  Coherence will be measured using Heart Rate Variability (HRV) biofeedback.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya, Petaling Jaya, WP KUALA LUMPUR, Malaysia

IPD SHARING:
Plan to Share IPD: No